CLINICAL TRIAL: NCT07122960
Title: Strengthening Informed Consent for Authentic Participation in Perinatal HIV Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Louise Kuhn, Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAV1833; 1R21HD115480 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Consent Form
Keywords: Consent process

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Informed Consent Form (ICF) (Experimental)
  Interventions: Other: Visual ICF
- Text-only Informed Consent Form (Active Comparator)
  Interventions: Other: Text-only ICF

INTERVENTIONS:
Other: Visual ICF — This visual ICF fully represents all the content of the standard, text-only ICF using cartoon characters, graphics and easy text.
  Arms: Visual Informed Consent Form (ICF)
Other: Text-only ICF — Text-only ICF
  Arms: Text-only Informed Consent Form

SUMMARY:
This study evaluates a visual Informed Consent Form (ICF) compared to a standard, text-only ICF as an approach to achieving meaningful consent into a clinical trial. The visual ICF uses cartoon characters, graphics and easy-to-understand text to cover the full content of a standard, text-only ICF. In this study, women who are considering enrollment into a clinical trial of a nutrition intervention for their infants will be randomized to either the visual ICF or to the text-only ICF. Qualitative and quantitative data will be collected immediately after the consent process and 8 weeks later. In addition, women not eligible for enrollment into the infant nutrition trial will be asked questions about their opinions regarding the visual ICF. The overall goal of the sub-study is to inform efforts to improve meaningful consent into clinical trials by evaluating whether the visual ICF improves understanding of the trial.

DETAILED DESCRIPTION:
The overall goal of the study is to inform efforts to improve meaningful consent into clinical trials. The investigators are evaluating whether substituting a visual informed consent form (ICF) for the usual text-only ICF will increase potential participants' understanding of the risks and benefits of research and contribute to more informed participation.

This study is nested within a larger clinical trial of a nutrition intervention for infants underway in South Africa. For this larger trial, a visual ICF was developed that covers the identical content of a standard text-only ICF. For this sub-study (n=40), women who are considering enrollment into this larger study who agree to enroll in the sub-study, will be randomized to either receive the visual ICF or to receive the text-only ICF. Following the decision to either participate or not in the larger trial, women will be interviewed about their knowledge recall of the content of the ICF including concerning the trial goal, the voluntary nature of participation, potential benefits, potential risks, and randomization measured using a mix of true/false/uncertain and likert-type response options. Questions will also be asked about decision conflict, self-rated understanding, self-efficacy, and satisfaction with the informed consent process. Eight weeks later, at one of the follow-up visits in the larger trial, these questions will be repeated to determine knowledge retention and decision regret and trust in the study team. The evaluation includes both quantitative and qualitative data which will be analyzed using standard mixed methods analysis techniques.

In addition, an independent population of women from the same area with infants of the same age but who are not eligible for the larger trial will be enrolled (n=20). For this population, participating in the trial is a hypothetical situation and thus respondents have no direct connection with the study team and thus are less prone to positive bias in responses. Questions will be asked concerning opinions about the visual ICF using a semi-structured, qualitative, think-aloud approach.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45 years of age
* Pregnant women or women that have recently given birth within the past 2-6 weeks

Exclusion Criteria:

* Unwilling to provide consent
* Severe maternal or infant illness (e.g. tuberculosis, major psychiatric or neurological conditions)
* Inability to communicate in one of the three languages (English, isiXhosa, or Afrikaans)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Summed score from the validated Quality of Informed Consent (QUIC) instrument. | Immediately after the consent process (Day 0) and 8 weeks later
  The QUIC measures knowledge recall. The summed score of 10 knowledge items comprising key concepts of informed consent will be calculated. The scores range between 0 and 22 with higher scores indicating higher knowledge.

SECONDARY OUTCOMES:
Self-rated Understanding | Immediately after consent process (Day 0)
  Six item self-rated assessment of understanding, which extends beyond knowledge recall to assess comprehension and ability to assimilate information. Scores range between 0-12 with higher scores indicating better understanding.
Decision Regret Scale | 8 weeks after consent process
  Validated measure with 5 items assessing attitudes about the decision making outcome. The possible score ranges are 0-10 with higher scores indicating less regret.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kuhn, PhD, Principal Investigator — Columbia University
Locations (1):
- Stellenbosch University Wooster Rural Campus, Worcester, Western Cape, South Africa